CLINICAL TRIAL: NCT06122402
Title: Effectiveness of Care Bundle in Preventing Medical Adhesive-Related Skin Injury Due to Central Venous Catheter Fixation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Özlem Şensoy, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUC-SENSOY-MARSI-001
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Skin Injury
Keywords: children; marsi; medical adhesive-related skin injury; care bundle; skin injury

STUDY DESIGN:
Intervention Model Description: The study is designed as a quasi-experimental study with a pre-test and post-test control group design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SECURE Care Bundle (Experimental): The SECURE Care Bundle has been developed by researchers based on the latest evidence to prevent medical adhesive-related skin injuries associated with central venous catheter fixation in children. The SECURE Care Bundle is a systematic approach to care that includes checking the skin, assessing risk factors, correctly applying and removing medical adhesives and registering medical adhesive related skin injury.
  Interventions: Other: SECURE Care Bundle
- Standart Care (Active Comparator): No intervention will be applied to this group. No intervention will be applied to this group. The care provided in the clinic will continue to be provided in the same way.
  Interventions: Procedure: Standart Care

INTERVENTIONS:
Other: SECURE Care Bundle — The SECURE Care Bundle is a systematic approach to care that includes checking the skin, assessing risk factors, registering medical adhesive related skin injury and correctly applying and removing medical adhesives including CHG dressing and silicone based remover.
  Arms: SECURE Care Bundle
Procedure: Standart Care — It is applied in routine care in the clinic. There is no standardization and no procedure for checking the skin, assessing risk factors, registering medical adhesive related skin injury and correctly applying and removing medical adhesives. Only CHG dressing is used for central venous catheter care.
  Arms: Standart Care

SUMMARY:
Skin injury due to the use of medical adhesives is a common but under recognized complication in children. To prevent central venous catheter-related complications, care interventions should be planned in such a way that they do not lead to medical adhesive-related skin injury. Systematic administration of preventive care interventions is needed to reduce skin injuries associated with medical adhesive used for central venous catheter fixation. The SECURE Care Bundle has been developed by researchers based on the latest evidence to prevent medical adhesive-related skin injuries associated with central venous catheter fixation in children.The SECURE Care Bundle is a systematic approach to care that includes checking the skin, assessing risk factors, correctly applying and removing medical adhesives and registering medical adhesive related skin injury.

This study aims to evaluate the effectiveness of the SECURE Care Bundle in reducing MARSI incidence related to CVC fixation in pediatric patients and to examine its influence on the MARSI occurrence time.

Hypotheses Null Hypothesis (H₀): There is no effect of the SECURE Care Bundle in preventing skin injuries related to central venous catheter (CVC) fixation in children.

Hypothesis 1 (H₁): Children who receive the SECURE Care Bundle experience a lower incidence of medical adhesive-related skin injury due to CVC fixation compared to those who receive standard care.

Hypothesis 2 (H₂): Children who receive the SECURE Care Bundle develop medical adhesive-related skin injury due to CVC fixation later than those who receive standard care.

This quasi-experimental study follows a pre-test/post-test control group design and will be conducted in the Pediatric Cardiovascular Intensive Care Unit. A total of 92 pediatric patients will participate. Following informed consent, patients will be allocated into intervention (n=46) and control (n=46) groups. Data collection tools will include a descriptive information form, the Braden QD Scale, a skin observation form, and the SECURE Care Bundle checklist. The intervention group will receive the SECURE Care Bundle, and its effectiveness will be assessed by analyzing MARSI incidence and time to onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 18 years.
* Underwent cardiovascular surgery and had a jugular central venous catheter (CVC) inserted.
* Admitted to the Pediatric Cardiovascular Intensive Care Unit (PCCU) in the postoperative period.
* Have a Braden QD Scale score of 12 or higher at admission.
* Parental informed consent obtained via a voluntary participation form.

Exclusion Criteria:

* Patients who had a central venous catheter inserted in another unit prior to cardiovascular surgery.
* Patients with pre-existing skin injury around the catheter site before insertion.
* Patients with a known history of dermatological disease.
* Patients with a known allergy to any of the products used in the study.
* Patients for whom catheter leakage occurs.
* Patients whose catheter is removed due to complications (e.g., infection, dislodgement, or other clinical reasons).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of medical adhesive-related skin injury due to central venous catheter fixation | From Day 1 (postoperative admission to PCCU) to MARSI occurrence or discharge, up to 30 days
  Incidence of medical adhesive-related skin injury due to central venous catheter fixation refers to the proportion of patients who develop medical adhesive-related skin injury (MARSI). This outcome will be assessed in both the pre-test and post-test groups, and the results will be compared to evaluate the effectiveness of the intervention.Three types of MARSI incidence rates will be calculated: (1)the rate per 100 patients, (2)the rate per 100 MAs, and (3)the rate per 1000 days of MA use. The formulas for calculating each incidence rate will be as follows: (1)incidence rate per 100 patients= number of MARSIs/number of patients × 100, (2)incidence rate per 100 MAs= number of MARSIs/number of MAs × 100, and (3)incidence rate per 1000 days of MA use= number of MARSIs/number of days of MA usage × 1000.

SECONDARY OUTCOMES:
MARSI occurrence time | From Day 1 (the day of CVC insertion and fixation) to the first occurrence of MARSI or end of treatment, up to 30 days
  MARSI occurrence time is defined as the time interval, measured in days, from the initial application of the central venous catheter (CVC) and its securement with medical adhesive to the first documented occurrence marsi.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Şensoy, Principal Investigator — İstanbul University-Cerrahpaşa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University- Cerrahpaşa, Istanbul, Şisli
  - Istanbul University- Cerrahpaşa, Istanbul, Şişli

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be become available upon request for three years.
Access Criteria: The data will become available upon request by contacting with principle investigator.

REFERENCES:
- [Derived] Sensoy O, Caglar S. SECURE Care Bundle to Prevent Medical Adhesive-Related Skin Injury in Paediatric Central Venous Catheter Fixation: A Study Protocol. Nurs Crit Care. 2025 Nov;30(6):e70226. doi: 10.1111/nicc.70226. PMID 41193400